CLINICAL TRIAL: NCT03690934
Title: Randomized Conrtolled Study: Fistula Laser Closure (FiLaC™) vs Monopolar Coagulation for Treatment of Complex Anal Fistulae.
Brief Title: Treatment of Transsphicteric Fistula-in-ano by Method of Laser Thermoobliteration(FiLaC™).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74
Record Dates: First submitted 2018-09-12; First posted 2018-10-01 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Intervention Model Description: Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fistula-tract laser closure (FiLAC™) (Experimental): The treatment technique consists of laser coagulation of fistulous tract walls with a diode laser with a wavelength of 1470 nm, which leads to thermo-obliteration of the fistulous tract.
  Interventions: Procedure: Fistula-tract laser closure (FiLAC™)
- Fistula monopolar cogulation (Active Comparator): The treatment technicque consists of monopolar coagulation of fistulous tract walls with suturing the internal fistulas opening.
  Interventions: Procedure: Monopolar coagulation of fistulous tract

INTERVENTIONS:
Procedure: Fistula-tract laser closure (FiLAC™) — The procedure was performed with a diode laser platform emitting laser energy of 15 W at a wavelength of 1470 nm by means of a radial ﬁber. For obliteration, the ﬁstula track is treated with a continuous slow retraction of the laser ﬁbre withdrawn at a rate of approximately 1 cm per 2-3s.
  Arms: Fistula-tract laser closure (FiLAC™)
Procedure: Monopolar coagulation of fistulous tract — The procedure was performed with a monopolar coagulator platform emitting monopolar coagulation. For obliteration, the ﬁstula track is treated with a continuous slow retraction of the monopolar energy with suturing the internal fistulas opening.
  Arms: Fistula monopolar cogulation

SUMMARY:
This is a randomized, controlled, parallel study to compare the results of treatment for patients with transsphincteric fistulas-in-ano.

DETAILED DESCRIPTION:
We are planning to eroll 120 patients in this study,the duration of the stady be 3 years. Each of two groups will include 60 people. Pationts in the first group will be assigned to get treatment of the fistula-in-ano by laser thermo-obliteration (FiLAC™), patietns of the second group will forego monopolar coagulation of the fistulas tract with suturing the internal fistulas opening.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent to the study;
2. Patients with high transsphincteric fistula (>1/3), suprasphincteric fistula whithout abscesses;
3. The presence of a formed fistulous tract > 2 cm in length.

Exclusion Criteria:

1. Suprasphincteric fistula with abscesses or infiltrates;
2. Extrasphincteric fistula;
3. Length of fistula tract < 2 cm;
4. The presence of sever scars in the region of internal fistula opening, wide fistula opening > 5 mm;
5. Crohn's fistulae

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of healing | 60 days
  healing

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia